CLINICAL TRIAL: NCT04339634
Title: Simulation of Risk of Adverse Drug Events Associated With the Initiation of Drugs Repurposed for the Treatment of COVID-19 in Frail Elderly Adults With Polypharmacy
Status: Completed | Type: Observational
Sponsor: Tabula Rasa HealthCare (Industry)
Responsible Party: Sponsor
Other Study IDs: COVID-PACE-2020-001
Record Dates: First submitted 2020-04-07; First posted 2020-04-09 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: COVID; Drug Effect; Drug Interaction; Adverse Drug Event
Keywords: COVID-19; Elderly; Adverse Drug Event; Repurposed Drug; Drug Interaction; LQTS
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Program of All-Inclusive Care for the Elderly: The Program of All-Inclusive Care for the Elderly (PACE) provides comprehensive medical and supportive services for community-dwelling persons, mostly older adults (>55 years), as an alternative to institutionalization. Medical services are provided by an interdisciplinary team of healthcare professionals, Tabula Rasa HealthCare being the pharmacy care provider for several PACE organizations.
  Interventions: Other: Simulation of Repurposed Drugs for COVID-19

INTERVENTIONS:
Other: Simulation of Repurposed Drugs for COVID-19 — This study is a simulation of adding repurposed drugs for COVID-19. We are using drug claims, and will not intervene with patient care.
  Other Names: Simulation using proprietary risk stratification software

SUMMARY:
This retrospective study aims to perform a medication risk stratification using drug claims data and to simulate the impact of the addition of various repurposed drugs on the Medication Risk Score (MRS) in elderly people enrolled in PACE organizations. Our clinical tool would enable to identify potential multi-drug interactions and potentially reduce the risk of adverse drug events (ADE) developing in elderly patients infected with COVID-19.

DETAILED DESCRIPTION:
Certain investigational agents have been described in observational series or are being used anecdotally based on in vitro or extrapolated evidence. It is important to acknowledge that there are no controlled data supporting the use of any of these agents, and their efficacy for COVID-19 is unknown. FDA-approved drugs such as chloroquine/hydroxychloroquine, lopinavir/ritonavir, monoclonal IL-6 antibodies, JAK inhibitors, thalidomide and the new investigational drug, remdesivir have been proposed for repurposing to fight COVID-19 and its complications.

A medication risk stratification strategy will be used to simulate the impacts of different potential repurposed drugs for COVID-19 on the Medication Risk Score (MRS) which is used as a predictive tool for ADEs. A retrospective study will be conducted using de-identified drug claims data of elderly patients with polypharmacy.

Patients meeting all the following criteria will be included:

1. Patient enrolled in a PACE organization during the implementation period;
2. PACE organization contractually receiving pharmacy services from CareKinesis;

Exclusion Criteria

a) No drug claims data available for the period of 2019-2020

This retrospective cohort will utilize 178,867 drug claims from approximately 12,123 patients enrolled in PACE. MRS will be calculated using the last available 3-month period of drug claims in 2019. The data elements required for the calculation of the full set of risk scores are: prescribed drugs, dose, age, gender. Medication risk stratification using 5 factors will be performed to obtain the MRS. Various repurposed drugs (drugs associated with the highest probability or efficacy or shown interest as per their inclusion in current clinical trials will be prioritized) will be added to the patient drug regimen except for the patients that are currently taking the repurposed drug. A new MRS will be generated for all stratified patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient enrolled in a PACE organization during the implementation period;
* PACE organization contractually receiving pharmacy services from CareKinesis;

Exclusion Criteria:

* No drug claims data available for the period of 2019-2020

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The Program of All-Inclusive Care for the Elderly (PACE) provides comprehensive medical and supportive services for community-dwelling persons, mostly older adults (>55 years), as an alternative to institutionalization. Medical services are provided by an interdisciplinary team of healthcare professionals, Tabula Rasa HealthCare being the pharmacy care provider for several PACE organizations.
Sampling Method: Non-Probability Sample
Enrollment: 12873 (Actual)
Dates: Start 2020-04-02 (Actual); Primary Completion 2023-01-30 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
To determine the Medication Risk Score of de-identified PACE's participants using their current drug regimen. | Three months
  Quantitative
To simulate the Medication Risk Score following the addition of different repurposed drugs against COVID-19 to their current drug regimen. | Three months
  Quantitative
To compare the impact on Medication Risk Score before and after the addition of repurposed drugs for COVID-19. | Three months
  Quantitative
To assess and compare the effects of various repurposed drugs for COVID-19 on each of the 5 factors computed by algorithms to derive the Medication Risk Score. | 3 months
  Quantitative

SECONDARY OUTCOMES:
To investigate the effects of various covariables on the Medication Risk Score in the presence of repurposed drugs for COVID-19. | 6 months
  Qualitative
To explore the effects on Medication Risk Score of various repurposed drugs for COVID-19 within subgroups of patients classified by specific diseases or drugs used. | 1 year
  Qualitative

CONTACTS AND LOCATIONS:
Overall Officials: Veronique Michaud, PhD, Principal Investigator — Tabula Rasa HealthCare
Locations (1):
- Tabula Rasa HealthCare Precision Pharmacotherapy Research and Development Institute, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Epidemiology Working Group for NCIP Epidemic Response, Chinese Center for Disease Control and Prevention. [The epidemiological characteristics of an outbreak of 2019 novel coronavirus diseases (COVID-19) in China]. Zhonghua Liu Xing Bing Xue Za Zhi. 2020 Feb 10;41(2):145-151. doi: 10.3760/cma.j.issn.0254-6450.2020.02.003. Chinese. PMID 32064853
- [Background] Hajjar ER, Cafiero AC, Hanlon JT. Polypharmacy in elderly patients. Am J Geriatr Pharmacother. 2007 Dec;5(4):345-51. doi: 10.1016/j.amjopharm.2007.12.002. PMID 18179993
- [Background] Mehta P, McAuley DF, Brown M, Sanchez E, Tattersall RS, Manson JJ; HLH Across Speciality Collaboration, UK. COVID-19: consider cytokine storm syndromes and immunosuppression. Lancet. 2020 Mar 28;395(10229):1033-1034. doi: 10.1016/S0140-6736(20)30628-0. Epub 2020 Mar 16. No abstract available. PMID 32192578
- [Background] Stabler T, Piette JC, Chevalier X, Marini-Portugal A, Kraus VB. Serum cytokine profiles in relapsing polychondritis suggest monocyte/macrophage activation. Arthritis Rheum. 2004 Nov;50(11):3663-7. doi: 10.1002/art.20613. PMID 15529362
- [Background] Vouri SM, Crist SM, Sutcliffe S, Austin S. Changes in Mood in New Enrollees at a Program of All-Inclusive Care for the Elderly. Consult Pharm. 2015 Aug;30(8):463-71. doi: 10.4140/TCP.n.2015.463. PMID 26260643
- See also: World Health Organization: COVID-19 — https://www.who.int/emergencies/diseases/novel-coronavirus-2019
- See also: Application of a Novel Medication-Related Risk Stratification — http://www.carekinesis.com/wp-content/uploads/2018_Cicali_B_Benefits_Q_Application_of_a_novel_medication-related_risk_stratification_strategy.pdf